CLINICAL TRIAL: NCT00001702
Title: Evaluation of the Association of Polymorphisms in the Innate Immune System With the Risk for Blastomycosis Dermatitidis Infection in Patients Not Infected With HIV and Complications Associated With Blastomycosis Dermatitidis Infection
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980138; 98-C-0138
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-10-06

CONDITIONS: Blastomycosis
Keywords: Genetic; Variant Alleles; Risk Factor; Cancer; Transplantation
MeSH Terms: conditions — Blastomycosis; Neoplasms

SUMMARY:
Innate immunity plays an important role for fungal recognition and initiation of fungicidal activity. We hypothesize that subtle differences in different molecules of innate immunity may contribute to either the predisposition or clinical course of infection with Blastomycosis dermatitidis. To test this hypothesis, we propose to analyze the allelic frequencies of 15 different genes (mannose binding lectin, Fc-gamma receptor IIa and IIb, Fc-gamma receptors IIIa and IIIb, myeloperoxidase, tumor necrosis factor-alpha and -beta, interleukin 1A and 1B, interleukin-1 receptor antagonist, interleukin-10, NRAMP-1, chitotriosidase, and chemokine receptor 5) and their intragenic polymorphic forms and to compare this data to the incidence and severity of Blastomycosis dermatitidis infection. With this study we hope to identify a group of molecules of innate immunity which influence the risk and severity of invasive Blastomycosis dermatitidis infection.

DETAILED DESCRIPTION:
Innate immunity plays an important role for fungal recognition and initiation of fungicidal activity. We hypothesize that subtle differences in different molecules of innate immunity may contribute to either the predisposition or clinical course of infection with Blastomycosis Dermatitidis. To test this hypothesis, we propose to analyze the allelic frequencies of 15 different genes (mannose binding lectin, Fc-gamma receptor Ila and IIb, Fc-gamma receptors IIIa and IIIb, myeloperoxidase, tumor necrosis factor-alpha and -beta, interleukin 1A and 1B, interleukin-1 receptor antagonist, interleukin-10, NRAMP-1, chitotriosidase, and chemokine receptor 5) and their intragenic polymorphic forms and to compare this data to the incidence and severity of Blastomycosis Dermatitidis infection. With this study we hope to identify a group of molecules of innate immunity which influence the risk and severity of invasive Blastomycosis Dermatitidis infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients in the database have been confirmed with a diagnosis of Blastomycosis dermatitides infection by a combination of isolation of the yeast form in a diagnostic microbiology laboratory and/or an elevated cryptococcal antigen titer (which is commercially available).

Only patients diagnosed and treated in the United States and Canada will be included in this analysis.

Only patients who are not co-infected with HIV will be included in the study.

Patient samples will be collected and clinical data will be evaluated only after signed consent has been obtained.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 1998-07-29; Primary Completion 2007-06-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Bellamy R, Ruwende C, Corrah T, McAdam KP, Whittle HC, Hill AV. Variations in the NRAMP1 gene and susceptibility to tuberculosis in West Africans. N Engl J Med. 1998 Mar 5;338(10):640-4. doi: 10.1056/NEJM199803053381002. PMID 9486992
- [Background] Blakemore AI, Tarlow JK, Cork MJ, Gordon C, Emery P, Duff GW. Interleukin-1 receptor antagonist gene polymorphism as a disease severity factor in systemic lupus erythematosus. Arthritis Rheum. 1994 Sep;37(9):1380-5. doi: 10.1002/art.1780370917. PMID 7945503
- [Background] Boot RG, Renkema GH, Strijland A, van Zonneveld AJ, Aerts JM. Cloning of a cDNA encoding chitotriosidase, a human chitinase produced by macrophages. J Biol Chem. 1995 Nov 3;270(44):26252-6. doi: 10.1074/jbc.270.44.26252. PMID 7592832